CLINICAL TRIAL: NCT01531933
Title: Phase III Clinical Study : DLBS3233 in Primary Prevention of Type 2 Diabetes Mellitus [DIPPER-DM]
Brief Title: Efficacy and Safety of DLBS3233 in Prediabetic Patients
Acronym: DIPPER-DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DLBS3233-0711
Record Dates: First submitted 2012-02-09; First posted 2012-02-13 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Prediabetic
Keywords: Prediabetic; Primary prevention; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — DLBS3233

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DLBS3233 (Experimental)
  Interventions: Drug: DLBS3233
- Placebo of DLBS3233 (Placebo Comparator)
  Interventions: Drug: Placebo of DLBS3233

INTERVENTIONS:
Drug: DLBS3233 — For the first 4 weeks, subjects should take DLBS3233 at the dose of 50 mg once daily. For the next (or last) 8 weeks, all subjects who do not respond well (poor responders) to the study regimen will receive a titrated dose of 100 mg once daily, while the (good) responders will remain at the previous dose regimen. Good responders are defined as those who achieve 2h-PG level of < 140 mg/dL or a decrease of 2h-PG level of ≥ 10% from baseline; otherwise will be called poor responders. At every study visit, subjects will be provided with an education on lifestyle modification given by the assigned nutritionist.
  Other Names: Inlacin
  Arms: DLBS3233
Drug: Placebo of DLBS3233 — For the first 4 weeks, subjects should take placebo of DLBS3233 at the dose of 50 mg once daily. For the next (or last) 8 weeks, all subjects who do not respond well (poor responders) to the study regimen will receive a titrated dose of 100 mg once daily, while the (good) responders will remain at the previous dose regimen. Good responders are defined as those who achieve 2h-PG level of < 140 mg/dL or a decrease of 2h-PG level of ≥ 10% from baseline; otherwise will be called poor responders. At every study visit, subjects will be provided with an education on lifestyle modification given by the assigned nutritionist.
  Arms: Placebo of DLBS3233

SUMMARY:
This is a 2-arm, prospective, double blind, randomized, and controlled clinical study for 12 weeks of therapy to investigate clinical efficacy and safety of DLBS3233.

It is hypothesized that DLBS3233 will delay the progress of beta-cell dysfunction as measured by the improvement of prandial (particularly the first phase) insulin secretion as well as insulin resistance in prediabetic subjects which may prevent the conversion of prediabetes into type 2 diabetes mellitus.

DETAILED DESCRIPTION:
There will be two groups of treatment in this study who will receive DLBS3233 or placebo of DLBS3233 for 12 weeks of therapy.

Subjects will be provided with an education on lifestyle modification given by the assigned nutritionist. All subjects will be advised to follow such a lifestyle modification throughout the study period.

All subjects will be under direct supervision of a medical doctor during the study period.

All clinical and laboratory examinations to evaluate the investigational drug's efficacy, will be performed at baseline, Week 8th and Week 12th (end) of study treatment. Blood glucose level (both FPG and 2h-PG) will be performed at baseline and at interval of 4 weeks over the 12 weeks of study treatment. Safety examinations will be performed at baseline and at the end of study. Occurrence of adverse event will be observed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with age of 18-60 years
* Prediabetic patients (2h-PPPG level of 140-199 mg/dL)
* Serum ALT ≤ 2.5 times upper limit of normal
* Serum creatinine < 1.5 times upper limit of normal
* Able to take oral medication

Exclusion Criteria:

* Female of childbearing potential
* History of diabetes mellitus
* History of symptomatic coronary arterial disease, stroke, and cardiovascular events
* Current treatment with systemic corticosteroids or herbal (alternative) medicines
* Any other disease state or uncontrolled illness, which judged by the investigator, could interfere with trial participation or trial evaluation
* Participation in any other clinical studies within 30 days prior to screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in 15-minute post prandial insulin level | 12 weeks of treatment
  Change in 15-minute post prandial insulin level from baseline to 12 weeks of treatment

SECONDARY OUTCOMES:
Change in 15-minute post prandial insulin level | 8 weeks of treatment
  Change in 15-minute post prandial insulin level from baseline to 8 weeks of treatment
Change in 2-hour post prandial insulin level | 8 weeks and 12 weeks of treatment
  Change in 2-hour post prandial insulin level from baseline to 8 weeks and to 12 weeks of treatment
Change in 15-minute post prandial plasma glucose | 8 weeks and 12 weeks of treatment
  Change in 15-minute post prandial plasma glucose from baseline to 8 weeks and to 12 weeks of treatment
Change in 2-hour post prandial plasma glucose | 4 weeks, 8 weeks, and 12 weeks of treatment
  Change in 2-hour post prandial plasma glucose from baseline to each study visit (4 weeks, 8 weeks, and 12 weeks of treatment)
Change in HOMA-IR | 8 weeks and 12 weeks of treatment
  Change in HOMA-IR from baseline to 8 weeks and to 12 weeks of treatment
Change in hs-CRP | 8 weeks and 12 weeks of treatment
  Change in hs-CRP from baseline to 8 weeks and to 12 weeks of treatment
Improvement in lipid profile | 8 weeks and 12 weeks of treatment
  Improvement in lipid profile from baseline to 8 weeks and to 12 weeks of treatment, including: fasting plasma HDL-cholesterol, fasting plasma triglyceride, 15-minute post prandial plasma triglyceride, and 2-hour post prandial plasma triglyceride
Change in adiponectin | 8 weeks and 12 weeks of treatment
  Change in adiponectin from baseline to 8 weeks and to 12 weeks of treatment
Change in waist-to-hip ratio | 4 weeks, 8 weeks, and 12 weeks of treatment
  Change in waist-to-hip ratio from baseline to each of study visit (4 weeks, 8 weeks, and 12 weeks of treatment)
ECG | 12 weeks of treatment
  ECG will be evaluated at baseline and at end of study (12 weeks of treatment)
Vital signs | 4 weeks, 8 weeks, and 12 weeks of treatment
  Vital signs (systolic and diastolic blood pressure, heart rate, respiration rate) will be evaluated at baseline and at each study visit (4 weeks, 8 weeks, and 12 weeks of treatment)
Body weight | 4 weeks, 8 weeks, and 12 weeks of treatment
  Body weight will be evaluated at baseline and at each study visit (4 weeks, 8 weeks, and 12 weeks of treatment)
Liver function | 12 weeks of treatment
  Liver function (levels of serum ALT, γ-GT, alkaline phosphatase) will be evaluated at baseline and at end of study (12 weeks of treatment)
Renal function | 12 weeks of treatment
  Renal function (serum creatinine level) will be evaluated at baseline and at end of study (12 weeks of treatment)
Adverse events | 1-12 weeks of treatment
  Adverse events as well as number of subjects experienced the events will be observed and evaluated during study period (12 weeks) and until all adverse events have been recovered or stabilized

CONTACTS AND LOCATIONS:
Overall Officials: Asman Manaf, Prof., Dr., dr., SpPD-KEMD, Principal Investigator — Department of Internal Medicine, dr. M. Djamil Padang Hospital
Locations (1):
- Department of Internal Medicine, dr. M. Djamil Padang Hospital, Padang, West Sumatera, Indonesia